CLINICAL TRIAL: NCT01457989
Title: Meta-Analysis of VRX-RET-E22-303 and VRX-RET-E22-304: Two Multicenter, Open-Label, Long-Term, Safety, Tolerability and Efficacy Studies of Retigabine in Adult Epilepsy Patients With Partial-onset Seizures (Extensions of Studies VRX-RET-E22-301 and VRX-RET-E22-302)
Brief Title: Meta-Analysis Plan for Pooled Data for Studies VRX-RET-E22-303 and VRX-RET-E22-304
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115476
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Epilepsy, Partial
Keywords: retention rate; epilepsy; responder rate; seizure freedom; discontinuation rate; safety assessment; reduction in seizure frequency; open-label
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — ezogabine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- retigabine/ezogabine: retigabine/ezogabine; dose range up to 1200 mg/day
  Interventions: Drug: retigabine/ezogabine

INTERVENTIONS:
Drug: retigabine/ezogabine — dose range up to 1200 mg/day
  Other Names: Trobalt

SUMMARY:
The objective of this meta-analysis is to provide data on long-term safety and efficacy following the recent positive Committee for Medicinal Products for Human Use (CHMP) opinion for retigabine using pooled data from ongoing open-label extension (OLE) Studies VRX-RET-E22-303 and VRX-RET-E22-304.

DETAILED DESCRIPTION:
Data from the October 2009 data-cut of ongoing Studies VRX-RET-E22-303 (Study 303) and VRX-RET-E22-304 (Study 304) will be pooled, summarized, and published with the goal of providing updated long-term safety and efficacy information for subjects and prescribers following the recent positive CHMP opinion for retigabine for adjunctive use in patients with partial seizures. Studies 303 and 304 are the open-label extensions of two Phase 3 studies (VRX-RET-E22-301 and VRX-RET-E22-302), respectively. Studies 301 and 302 were randomized, double-blind, placebo-controlled, parallel-group, multicenter studies of 600 mg and 900 mg per day (Study 302) and 1200 mg per day (Study 301). All subjects who wished to enter the OLE studies and, in the opinion of the investigator, were expected to benefit from participation in the OLEs, entered a 6-week (Study 301) or 4-week (Study 302) transition phase in which their dose of retigabine was titrated to or maintained at 400 mg TID (Study 301) or 300 mg TID (Study 302). Upon completion of the Transition phase, subjects enrolled into the extension studies. Once enrolled in the OLE, doses could be adjusted within the range of 600 mg to 1200 mg per day. Treatment in Studies 303 and 304 is planned to continue until regulatory approval and commercialization of retigabine or until the program is discontinued.

ELIGIBILITY:
This is meta-analysis therefore Inclusion/Exclusion criteria are not applicable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with partial onset seizures who have successfully completed the transition phase of VRX-RET-E22-301 and VRX-RET-E22-302.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | during open-label drug exposure up to database cutoff (max 40 months)
  Adverse events were the primary means to assess safety.

SECONDARY OUTCOMES:
Time to Discontinuation | during open-label extension up to date of discontinuation; subjects who continue in the study are censored at database cutoff (max 40 months)
  Time to discontinuation in number of days since first dose in open-label extension until subject discontinues
The number and percent of subjects exposed to study drug | for at least 3, 6, 12, 18, 24 and 32 months
  The number and percent of subjects exposed to study drug
Listing of abnormal liver function test results and liver adverse events | during open-label drug exposure up to database cutoff (max 40 months)
  Abnormal lab results if reported as adverse events or values of alkaline phosphatase, alanine transaminase, aspartate transaminase [>3, >5, >10xupper limit of normal (ULN)] or total bilirubin (>1.5, >2, >4xULN); treatment emergent adverse events related to liver function test abnormalities
Observed values and change from baseline summaries for American Urological Association symptom index scores, Post-Void Residual bladder ultrasound, Vital Signs and Weight | baseline (parent study) and at 1, 3, 12, 24 and 36 months
  Univariate statistics summarizing the observed values and change from baseline, using parent study baseline value
Percent change from baseline in seizure frequency | entire open-label extension period up to database cutoff (max 40 months)
  Percent change from baseline in 28-day total partial seizure frequency, using parent study baseline value.
Number and percent of responders | entire open-label extension period up to database cutoff (max 40 months)
  Number and percent of responders (defined as subjects with >=50% reduction from baseline in 28-day total partial seizure frequency) using parent study baseline value
Number and percent of seizure free subjects | during open-label drug exposure up to database cutoff (max 40 months)
  Percent of subjects seizure free for any 6 continuous months or longer for subjects treated for at least 6, 12 and 24 months; percent of seizure free subjects for any 12 continuous months or longer for subjects treated for at least 12 and 24 months
Proportion of subjects retained in the study | at 3, 6, 12, 24 and 32 months after exposure to first dose in open-label extension study.
  Length of time subjects retained in OLE as summarized by proportion of subjects remaining in both studies at given timepoints.
Mean of average dose | entire open-label drug extension period up to database cutoff (max 40 months)
  Mean average dose for all subjects combined and by modal dose category [the range of doses (<=750 mg/day, >750 to 1050 mg/day, >1050 mg/day) taken most frequently].

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline